CLINICAL TRIAL: NCT06422741
Title: Effect of a Grape Seed Proanthocyanidin Extract (GSPE) on LDL Cholesterol Levels in Rotating Night Shift Workers With Moderate Hypercholesterolemia. Randomized, Crossover, Controlled and Triple Blind Study.(CIRCAFENOL)
Brief Title: Effect of a Grape Seed Proanthocyanidin Extract (GSPE) on LDL Cholesterol Levels in Rotating Night Shift Workers
Acronym: CIRCAFENOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Eurecat (Other)
Collaborators: University Rovira i Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIRCAFENOL
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Circadian Rhythm Sleep Disorder, Shift Work Type; Cholesterol Level, High
Keywords: Proanthocyanidins; Circadian Rhythm; Metabolic Syndrome; Melatonin; Polyphenols
MeSH Terms: conditions — Cardiovascular Diseases; Sleep Disorders, Circadian Rhythm; Hypercholesterolemia; Metabolic Syndrome | interventions — Grape Seed Proanthocyanidins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- grape seed proanthocyanidin extract (Experimental): Participants will receive the grape seed proanthocyanidin extract (GSPE) for 6 weeks.
  Interventions: Dietary Supplement: grape seed proanthocyanidin extract
- Placebo (Placebo Comparator): Participants will receive the placebo for 6 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: grape seed proanthocyanidin extract — 250 mg of product presented in capsule form will be given.
  Arms: grape seed proanthocyanidin extract
Dietary Supplement: Placebo — 165 mg of cellulose will be given presented in capsule form.
  Arms: Placebo

SUMMARY:
The physiological processes of the body present daily oscillations called circadian rhythm. The circadian rhythm is essential for maintaining the vital functions of organisms, intervening directly and indirectly in a multitude of key processes, such as hormone secretion, cycles of activity and rest throughout the day, body temperature, the metabolism or absorption, processing and detoxification of nutrients. There are factors such as certain work schedules, prolonged exposure to screens, certain eating patterns or social jetlag, which have a negative impact on the circadian rhythm, causing its disruption and favoring the appearance of health alterations. Thus, there is evidence that associates night shift work with a higher incidence of risk factors for developing metabolic syndrome and cardiovascular diseases, including obesity, elevated blood levels of glucose, triglycerides, and low-density lipoprotein cholesterol (LDL-C), as well as lower levels of high-density lipoprotein cholesterol (HDL-C). In addition, disorders in the sleep cycle are associated with the development of hypertension and type 2 diabetes.

Several previous studies show that a grape seed proanthocyanidin extract (GSPE) has beneficial effects on different parameters by restoring the circadian rhythm.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the effect of daily GSPE intake, in combined with dietary recommendations, on LDL-C levels in individuals with rotating night shift work.

The secondary objectives are to evaluate the effects of GSPE on: anthropometric parameters,blood pressure, heart rate and endothelial function, markers of lipid and carbohydrate metabolism and insulin resistance, atherogenic indices, circulating levels of sex hormones and those related to hunger, satiety and stress; markers of systemic inflammation; circadian rhythm markers and sleep quality; level of physical activity, energy consumption, and changes in gene expression of key metabolic enzymes.

A randomized, crossover, placebo-controlled, triple-blind nutritional intervention study will be conducted. The study will be carried out in a population of 22 volunteers. Men and women aged 18 years or older, who are working a rotating night shift for at least 1 year and with blood levels of LDL-C between 116 and 190 mg/dL may participate.

Each volunteer will make 5 visits to the facilities of the EURECAT Nutrition and Health Technological Unit, in accordance with the study design:

* A pre-selection visit (to check inclusion/exclusion criteria), and if the inclusion criteria are met.
* Two study visits during consumption of the first product (GSPE or placebo), which will take place on the first day of study (visit 1) and after 6 weeks of treatment (visit 2).
* Two study visits during consumption of the second product (GSPE or placebo), which will take place after a three-week washout period (visit 3), and after 6 weeks of treatment (visit 4).

The main variable of the CIRCAFENOL study is circulating LDL-C levels.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years or older.
* Follow a rotating night shift work schedule* for at least one year before the start of the study.

  * shift workers with at least 5 night shifts per month alternating with day and/or afternoon shifts, with a seniority equal to or greater than one year.
* Have no intention of changing the work shift during the course of the study.
* Circulating LDL-C levels between 116 -190 mg/dL*, without pharmacological treatment with antihypertensives and/or lipid-lowering agents.

  *Values of 116 to 190 mg/dl indicate moderate alteration in the lipid profile and a greater risk of suffering from cardiovascular diseases, according to the European Society of Cardiology, and the European Society of Atherosclerosis.
* Have signed the informed consent before starting the study.
* Know how to read, write and speak in Catalan or Spanish

Exclusion Criteria:

* BMI values > 30 kg/m2
* Take supplements, multivitamin supplements (Vit.D, Vit. E and Vit.C), mineral supplements (Zinc, Selenium), essential fatty acids (omega-3), polyphenols, natural plant extracts, or phytotherapeutic products that interfere with the treatment under study.
* Consumption of alcoholic beverages:

  * Men: consume 4 or more Standard Beverage Units daily or 28 Standard Beverage Units weekly.
  * Women: Consume 2 or more Standard Beverage Units daily or 17 Standard Beverage Units weekly.
* Be an active smoker.
* Having lost more than 3 kg of weight in the last 3 months.
* Present food intolerances and/or allergies related to the study products, such as hypersensitivity to cellulose or proanthocyanidins.
* Present any chronic or autoimmune disease in clinical manifestation that may affect the results of the study such as diabetes (type I or II), cardiovascular disease, chronic kidney disease, hyper or hypothyroidism, chronic gastrointestinal diseases or cancer.
* Present familial hypercholesterolemia.
* Present hypertension (Systolic ≥140 mmHg; Diastolic ≥90 mmHg)
* Present any previous cardiovascular disease defined as myocardial infarction, angina pectoris, stroke or peripheral arterial disease.
* Individuals with treatment in the last 3 months before the start of the study with lipid-lowering, antidiabetic and/or antihypertensive drugs, or other drugs that may interfere with the results of the study.
* Taking supplements with polyphenol components or those aimed at lipid or blood pressure control in the last 3 months before the start of the study or during participation in the study.
* Follow a diet to lose weight, or very restrictive types of eating, such as intermittent fasting, ketogenic diet, etc.
* Being pregnant or intending to become pregnant.
* Being breastfeeding.
* Be participating or have participated in a clinical trial with medications or nutritional intervention study in the last 30 days before inclusion in the study.
* Suffering from eating disorders or psychiatric disorders.
* Being unable to follow study guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in LDL cholesterol levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum LDL cholesterol levels will be measured by commercial colorimetric kit.

SECONDARY OUTCOMES:
Change in body weight. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Body weight will be measured by standardized method.
Height. | At week 1.
  Height will be measured by standardized method.
Change in BMI. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Weight and height will be combined to report BMI in kg/m^2.
Change in waist circumference. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Waist circumference will be measured using a measuring tape.
Change in conicity index. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Weight, height and waist circumference will be combined to report Conicity index.
Change in waist circumference to height ratio. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Waist circumference and height will be combined to report Waist circumference to Height ratio.
Change in the amount of body fat. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Body fat will be measured by TANITA SC330.
Change in the amount of muscle mass. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Muscle mass will be measured by TANITA SC330.
Change in the amount of bone mass. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Bone mass will be measured by TANITA SC330.
Change in the amount of total body water. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Total body water will be measured by TANITA SC330.
Change in systolic blood pressure. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Systolic blood pressure will be measured using an automatic sphygmomanometer.
Change in diastolic blood pressure. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Diastolic blood pressure will be measured using an automatic sphygmomanometer.
Change in resting heart rate. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Resting heart rate will be measured using an automatic sphygmomanometer.
Change in endothelial function. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Endothelial function will be measured using the Laser-Doppler technique.
Change in serum total cholesterol levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum total cholesterol levels will be measured by standardized ultraviolet-visible spectrophotometry methods.
Change in serum HDL-c levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum HDL-c levels will be measured by standardized ultraviolet-visible spectrophotometry methods.
Change in serum Triglycerides levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum triglycerides levels will be measured by standardized ultraviolet-visible spectrophotometry methods.
Change in total cholesterol to HDL-c ratio. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Total cholesterol and HDL-c values will be combined to report Total cholesterol to HDL-c ratio.
Change in LDL-c to HDL-c ratio. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  LDL-c and HDL-c values will be combined to report LDL-c to HDL-c ratio.
Change in Plasma atherogenic index. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Plasma atherogenic index will be calculated as the logarithm of the triglycerides levels to HDL-c levels ratio.
Change in serum glucose levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum glucose levels will be measured by standardized ultraviolet-visible spectrophotometry methods.
Change in serum insulin levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum insulin levels will be measured by spectrophotometry methods.
Change in serum glycosylated hemoglobin levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum glycosylated hemoglobin levels will be measured by commercial kits.
Change in Homeostatic Model Assessment from Insulin Resistance Index (HOMA-IR). | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  HOMA-IR will be calculated using serum glucose and insulin levels.
Change in serum high sensitivity c-reactive protein levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum C-Reactive protein levels will be measured by plate test and by the agglutination of latex particles.
Change in serum ghrelin levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum ghrelin levels will be measured by ELISA kits.
Change in serum leptin levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum leptin levels will be measured by ELISA kits.
Change in circulating thyroid hormone T3 levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum T3 levels will be measured by liquid chromatography coupled to mass spectrometry with triple quadrupole detector (LC-TQD-MS/MS).
Change in circulating thyroid hormone T4 levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  SerumT4 levels will be measured by liquid chromatography coupled to mass spectrometry with triple quadrupole detector (LC-TQD-MS/MS).
Change in circulating testosterone levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum testosterone levels will be measured by liquid chromatography coupled to mass spectrometry with triple quadrupole detector (LC-TQD-MS/MS).
Change in circulating estrone levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum estrone levels will be measured by liquid chromatography coupled to mass spectrometry with triple quadrupole detector (LC-TQD-MS/MS).
Change in circulating 17-β-Estradiol levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum 17-β-Estradiol levels will be measured by liquid chromatography coupled to mass spectrometry with triple quadrupole detector (LC-TQD-MS/MS).
Change in circulating estriol levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum estriol levels will be measured by liquid chromatography coupled to mass spectrometry with triple quadrupole detector (LC-TQD-MS/MS).
Change in serum melatonin levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Serum melatonin levels will be measured by liquid chromatography coupled to mass spectrometry with triple quadrupole detector (LC-TQD-MS/MS).
Change in urine 6-Sulfatoxymelatonin levels. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  6-Sulfatoxymelatonin levels will be measured in spontaneous urine samples from two times of the day: morning and night by ELISA kit.
Change in activity and rest cycles (subjective measurement). | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Activity and rest cycles will be measured subjectively by dream diaries.
  The sleep diary will be self-completed by the participant and will determine the time at which the person attempted to sleep, the duration and interruptions of nighttime sleep, the person's sleep pattern, and how much of the day the person was active.
Change in activity and rest cycles (objective measurement). | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Activity and rest cycles will be measured objectively by actigraphs.
  The wrist actigraphs will be worn 24 hours a day and will measure heart rate, which will give an idea of the amount of time the person was asleep and active.
Pittsburgh Sleep Quality Index. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  It is a validated scale that measures the usual sleep habits during the past month. It consist of 7 areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. It contains a total of 19 items, grouped into 10 questions where each of the areas evaluated is a scored between 0 and 3. The scores from the seven areas are finally added up to give an overall score. The component score are summed to produce a global score (range 0 to 21). Higher score indicate worse sleep quality.
Chronotype. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  The chronotype will be evaluated using the Horne-Ostberg Morningness-Eveningness Questionnaire. Which consists of 19 questions that will allow volunteers to be classified into morning, night or intermediate people.
Change in circulating GSPE metabolites. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  GSPE metabolites will be measured by LC-TQD-MS/MS.
Change in food consumption habits. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Food consumption will be evaluated through a 3-day food record.
Change in Physical activity. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Physical activity will be evaluated through the Physical Activity Questionnaire, Quick Physical Activity Classifier, adapted from the PEFS guide of the Generalitat de Catalunya. The questionnaire asks about three specific types of activity (walking, moderate-intensity activities and vigorous intensity activities) in the set domains leisure time, domestic and gardening (yard) activities, work-related and transport-related activities. Frequency and duration are collected separately for each specific type of activity.
Change in body temperature. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Body temperature will be measured using a infrared thermometer according to a standardized measurement protocol.
Change in gene expression in peripheral blood mononuclear cells. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  The expression of key genes in lipid and carbohydrate metabolism and regulation of the circadian rhythm will be measured through transcriptomic analysis, performing RNA extraction, conversion to cDNA and subsequent analysis.
Change in serum metabolite profile. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  serum metabolites will be determined by LC-TQD-MS/MS.
Adverse events | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Possible adverse events derived from taking study's products will be recorded.
Consumption of dietary supplements. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Dietary supplements consumed during the study will be recorded in the case report form.
Concomitant medication. | Before (baseline) and after treatment period (6 weeks) for each of the two treatments (GSPE and placebo).
  Concomitant medication will be recorded in the case report form.
Age. | At week 1.
  Age will be recorded in years. It will be recorded in the case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Caimari Palou, PhD, Principal Investigator — UTNS (Eurecat, Reus)
Locations (2):
- Spain (2):
  - Eurecat, Reus, Tarragona
  - Fundació EURECAT, Reus, Tarragona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Technological Centre of Nutrition and Health. Eurecat_Reus — http://eurecat.org